CLINICAL TRIAL: NCT06647719
Title: Patient Directed Care After Carpal Tunnel Release Using Video Integration and Digital Education After Operations (VIDEO)
Brief Title: Postoperative Care After Carpal Tunnel Release Using Short Educational Videos
Acronym: VIDEO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Principal Investigator, Cesar J Bravo, Orthopedic Hand and Upper Extremity Surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-1469
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Carpal Tunnel Syndrome; Patient Satisfaction
Keywords: Carpal tunnel release (CTR); Patient-directed care; Educational videos; Minor hand surgery
MeSH Terms: conditions — Carpal Tunnel Syndrome; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): In-person group will be followed with standard -of-care postoperative clinic visits with a hand & upper extremity orthopaedic surgeon at Carilion Clinic Institute for Orthopaedics and Neurosciences at 2 weeks and 6 weeks from date of service.
- Video Management (Experimental): Postoperative education will be provided with 3 short videos that will be accessible to patients on all social media platforms and through MyChart with no scheduled in person postoperative visits. Patients will have a one time visit with either nurse or orthopaedic technician for suture removal 10-14 days from surgery if the participant has nonabsorbable sutures placed during surgery.
  Interventions: Other: Educational Videos

INTERVENTIONS:
Other: Educational Videos — Subjects in the experimental group will be provided with 3 links to videos to be watched after CTR surgery. These videos will be available through YouTube, Twitter, Facebook, Instagram, TikTok, or MyChart. Videos will be available to watch multiple times at the subjects choice.
  Arms: Video Management

SUMMARY:
The goal of this clinical trial is to learn if a patient-directed postoperative care program, using short educational videos, can improve patient satisfaction and reduce healthcare resource utilization in patients undergoing carpal tunnel release (CTR). The main questions it aims to answer are:

Will patients in the video-based care program be more satisfied with their postoperative care? Will this approach reduce healthcare resource use and the burden on patients without increasing complication rates? Researchers will compare the video-based patient-directed care group to the standard in-person follow-up group to see if patient satisfaction and resource use differ while maintaining similar outcomes and complication rates.

Participants will:

Watch three short educational videos (< 60 seconds each) on postoperative care. Schedule a suture removal appointment with a nurse at their convenience if needed.

Continue to have access to their provider through traditional methods such as phone, EMR, or urgent in-person visits.

DETAILED DESCRIPTION:
Carpal tunnel release (CTR) is a commonly performed procedure with predictable outcomes and a low complication rate. Traditionally, patients are scheduled for two postoperative follow-up visits-one at two weeks and another at six weeks. However, these routine visits rarely lead to a change in patient management and often impose logistical and financial burdens on patients, particularly for those living in rural areas who must travel long distances to their healthcare provider's clinic.

This study proposes an alternative postoperative care model for CTR patients that leverages short educational videos and allows patients to manage their recovery more independently. The experimental group in the study will receive three brief (< 60 seconds each) educational videos after surgery. These videos will cover key aspects of postoperative care, including wound management and when to seek medical attention. Unlike the traditional model, patients in this group will not have scheduled in-person or virtual follow-up visits unless they require them. All patients in the experimental group will still have access to their healthcare provider through standard communication channels, such as:

Calling the office for advice or concerns. Sending secure messages through the electronic medical record (EMR) system. Attending urgent in-person visits if necessary. If nonabsorbable sutures are used during surgery, patients in the experimental group will schedule an appointment for suture removal with a nurse at their convenience, usually 10-14 days post-surgery.

The primary goal of the study is to determine whether this patient-directed care model, which utilizes educational videos, can improve patient satisfaction and reduce the use of healthcare resources without compromising care quality or increasing complication rates.

Specific Aim: The study aims to evaluate whether a patient-directed postoperative care program for CTR can:

Improve patient satisfaction. Reduce healthcare resource utilization. Lessen the burden of care (e.g., fewer missed workdays and less time spent on healthcare-related activities).

Maintain comparable patient-reported outcomes, complication rates, and the number of urgent visits as those observed in traditional in-person follow-up care.

Hypotheses:

Patients who receive the educational videos will report higher satisfaction with their care.

These patients will miss fewer days of work and spend less time on health-related activities.

The experimental group will consume fewer healthcare resources (e.g., fewer clinic visits).

Patient-reported outcomes, complication rates, and urgent visits will be similar between the experimental and standard in-person care groups.

Significance: The results of this study have the potential to transform and enhance postoperative care for patients undergoing CTR and other minor surgical procedures. By reducing the need for routine in-person visits, the proposed care model can help alleviate the burden on patients, particularly those from rural areas. Additionally, reducing clinic utilization for straightforward postoperative cases could increase the availability of clinic appointments for more complex cases, thereby improving overall healthcare system efficiency. This patient-directed model could also be expanded to other surgical and nonsurgical conditions, empowering patients to take a more active role in their recovery while maintaining high standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either endoscopic (CPT 29848) or open CTR (CPT 64721)
* Access to a smartphone, tablet, or computer to view educational videos
* Access to internet to download or view postoperative education videos
* Age 18 or older

Exclusion Criteria:

* Patients undergoing any additional procedures
* Worker's compensation status
* Revision procedures
* Patients unable to utilize technology to view videos or follow instructions
* Patients with no access to internet
* Inability to provide informed consent for the study
* Patients unable to speak English fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) / Upper Extremity Computer Adaptive Test (UE CAT) / 5-Point Likert Scale | 2 and 6 weeks postoperatively
  All patient reported outcome measures will be reported at 2 and 6 weeks postoperatively. All responses will be recorded within the study's REDCap data base.

SECONDARY OUTCOMES:
Time Taken Off Work | Baseline to 6 week follow up
  Reported by patient or care giver during 2 and 6-week postoperative visits. (hours)
Travel time. | Baseline to 6 week follow up
  Time spent traveling to attend postoperative care appointments. (hours)
Number of Unplanned Visits | Baseline to 6 week follow up.
  The number of visits that were not originally scheduled as a part of standard of care procedures.
Patient Satisfaction Questionnaire | Baseline to 6 week follow up.
  Will record patient satisfaction as well as the number of unplanned visits, time taken off of work (hours), and travel time to attend appointments for postoperative care (hours).
Wound Complications | Baseline to 6 week follow up.
  Electronic Medical Records review will be performed to determine: Number of wound complications.
Total In Person Postoperative Visits | Baseline to 6 week follow up.
  Electronic Medical Records review will be performed to determine: Total number of in person postoperative visits

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Bravo, M.D., Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic Orthopaedic Surgery, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenfield PT, Manz WJ, DeMaio EL, Duddleston SH, Xerogeanes JW, Scott Maughon T, Spencer CC, Dawes A, Boden SD, Hammond KE, Wagner ER, Gottschalk MB, Daly CA, Pombo MW. Telehealth Can Be Implemented Across a Musculoskeletal Service Line Without Compromising Patient Satisfaction. HSS J. 2021 Feb;17(1):36-45. doi: 10.1177/1556331620977171. Epub 2021 Feb 21. PMID 33967640
- [Background] https://www. pewresearch.org/internet/fact-sheet/social-media/?menuItem=81867c91- 92ad-45b8-a964-a2a894f873ef
- [Background] Kim SH, Koh WU, Rhim JH, Karm MH, Yu HS, Lee BY, Shin JW, Leem JG. Preconsent video-assisted instruction improves the comprehension and satisfaction in elderly patient visiting pain clinic. Korean J Pain. 2012 Oct;25(4):254-7. doi: 10.3344/kjp.2012.25.4.254. Epub 2012 Oct 4. PMID 23091686
- [Background] Denny MC, Vahidy F, Vu KY, Sharrief AZ, Savitz SI. Video-based educational intervention associated with improved stroke literacy, self-efficacy, and patient satisfaction. PLoS One. 2017 Mar 23;12(3):e0171952. doi: 10.1371/journal.pone.0171952. eCollection 2017. PMID 28333925
- [Background] Kim S, Ju MK, Son S, Jun S, Lee SY, Han CS. Development of video-based educational materials for kidney-transplant patients. PLoS One. 2020 Aug 3;15(8):e0236750. doi: 10.1371/journal.pone.0236750. eCollection 2020. PMID 32745145
- [Background] Veldhuijzen G, Klemt-Kropp M, Terhaar Sive Droste JS, van Balkom B, van Esch AAJ, Drenth JPH. Computer-based patient education is non-inferior to nurse counselling prior to colonoscopy: a multicenter randomized controlled trial. Endoscopy. 2021 Mar;53(3):254-263. doi: 10.1055/a-1225-8708. Epub 2020 Nov 5. PMID 32702759
- [Background] Kuba MHM, Izuka BH. One Brace: One Visit: Treatment of Pediatric Distal Radius Buckle Fractures With a Removable Wrist Brace and No Follow-up Visit. J Pediatr Orthop. 2018 Jul;38(6):e338-e342. doi: 10.1097/BPO.0000000000001169. PMID 29529004
- [Background] Gamble D, Jenkins PJ, Edge MJ, Gilmour A, Anthony IC, Nugent M, Rymaszewski LA. Satisfaction and functional outcome with "self-care" for the management of fifth metacarpal fractures. Hand (N Y). 2015 Dec;10(4):607-12. doi: 10.1007/s11552-015-9749-8. Epub 2015 Feb 18. PMID 26568712
- [Background] Vusirikala A, Ensor D, Asokan AK, Lee AJ, Ray R, Tsekes D, Edwin J. Hello, can you hear me? Orthopaedic clinic telephone consultations in the COVID-19 era- a patient and clinician perspective. World J Orthop. 2021 Jan 18;12(1):24-34. doi: 10.5312/wjo.v12.i1.24. eCollection 2021 Jan 18. PMID 33520679
- [Background] Orrange S, Patel A, Mack WJ, Cassetta J. Patient Satisfaction and Trust in Telemedicine During the COVID-19 Pandemic: Retrospective Observational Study. JMIR Hum Factors. 2021 Apr 22;8(2):e28589. doi: 10.2196/28589. PMID 33822736
- [Background] Reider-Demer M, Raja P, Martin N, Schwinger M, Babayan D. Prospective and retrospective study of videoconference telemedicine follow-up after elective neurosurgery: results of a pilot program. Neurosurg Rev. 2018 Apr;41(2):497-501. doi: 10.1007/s10143-017-0878-0. Epub 2017 Jul 22. PMID 28735437
- [Background] Kane LT, Thakar O, Jamgochian G, Lazarus MD, Abboud JA, Namdari S, Horneff JG. The role of telehealth as a platform for postoperative visits following rotator cuff repair: a prospective, randomized controlled trial. J Shoulder Elbow Surg. 2020 Apr;29(4):775-783. doi: 10.1016/j.jse.2019.12.004. PMID 32197766
- [Background] Williams M, Amin A, Getgood A, Hallam P, Chojnowski AJ, Chapman PG. Telephone clinic follow-up following carpal tunnel decompression. J Hand Surg Eur Vol. 2008 Oct;33(5):641-4. doi: 10.1177/1753193408090124. Epub 2008 Jun 25. PMID 18579622
- [Background] Grandizio LC, Mettler AW, Caselli ME, Pavis EJ. Telemedicine After Upper Extremity Surgery: A Prospective Study of Program Implementation. J Hand Surg Am. 2020 Sep;45(9):795-801. doi: 10.1016/j.jhsa.2020.06.002. Epub 2020 Jul 18. PMID 32693989
- [Background] Kummerow Broman K, Roumie CL, Stewart MK, Castellanos JA, Tarpley JL, Dittus RS, Pierce RA. Implementation of a Telephone Postoperative Clinic in an Integrated Health System. J Am Coll Surg. 2016 Oct;223(4):644-51. doi: 10.1016/j.jamcollsurg.2016.07.010. Epub 2016 Aug 18. PMID 27545100
- [Background] Parisien RL, Shin M, Constant M, Saltzman BM, Li X, Levine WN, Trofa DP. Telehealth Utilization in Response to the Novel Coronavirus (COVID-19) Pandemic in Orthopaedic Surgery. J Am Acad Orthop Surg. 2020 Jun 1;28(11):e487-e492. doi: 10.5435/JAAOS-D-20-00339. PMID 32459409
- [Background] https://www.pewresearch.org/internet/fact-sheet/mobile/
- [Background] Rizzi AM, Polachek WS, Dulas M, Strelzow JA, Hynes KK. The new 'normal': Rapid adoption of telemedicine in orthopaedics during the COVID-19 pandemic. Injury. 2020 Dec;51(12):2816-2821. doi: 10.1016/j.injury.2020.09.009. Epub 2020 Sep 16. PMID 32951916
- [Background] Sultan AA, Acuna AJ, Samuel LT, Rabin JM, Grits D, Gurd DP, Kuivila TE, Goodwin RC. Utilization of Telemedicine Virtual Visits in Pediatric Spinal Deformity Patients: A Comparison of Feasibility and Patient Satisfaction at a Large Academic Center. J Pediatr Orthop. 2020 Sep;40(8):e712-e715. doi: 10.1097/BPO.0000000000001553. PMID 32235192
- [Background] Halonen LM, Vasara H, Stenroos A, Kosola J. Routine follow-up is unnecessary after intramedullary fixation of trochanteric femoral fractures-Analysis of 995 cases. Injury. 2020 Jun;51(6):1343-1345. doi: 10.1016/j.injury.2020.03.033. Epub 2020 Mar 10. PMID 32220506
- [Background] Tofte JN, Anthony CA, Polgreen PM, Buckwalter JA, Caldwell LS, Fowler TP, Ebinger T, Hanley JM, Dowdle SB, Holte AJ, Arpey NC, Lawler EA. Postoperative care via smartphone following carpal tunnel release. J Telemed Telecare. 2020 May;26(4):223-231. doi: 10.1177/1357633X18807606. Epub 2018 Nov 14. PMID 30428766
- [Background] Zhang D, Blazar P, Earp BE. Rates of Complications and Secondary Surgeries of Mini-Open Carpal Tunnel Release. Hand (N Y). 2019 Jul;14(4):471-476. doi: 10.1177/1558944718765226. Epub 2018 Mar 20. PMID 29557679
- [Background] Matsis R, Chou J, Clode N. Outcome of carpal tunnel decompression with pre-surgical diagnosis determined on general practitioner assessment and nerve conduction study. J Clin Orthop Trauma. 2020 Sep 6;13:15-18. doi: 10.1016/j.jcot.2020.08.028. eCollection 2021 Feb. PMID 33717870
- [Background] Sun Cao P, Loewenstein SN, Timsina LR, Adkinson JM. The Association of Insurance Status and Complications After Carpal Tunnel Release. Hand (N Y). 2023 Mar;18(2):192-197. doi: 10.1177/1558944721990818. Epub 2021 Feb 25. PMID 33631982
- [Background] Fajardo M, Kim SH, Szabo RM. Incidence of carpal tunnel release: trends and implications within the United States ambulatory care setting. J Hand Surg Am. 2012 Aug;37(8):1599-605. doi: 10.1016/j.jhsa.2012.04.035. Epub 2012 Jun 23. PMID 22727925
- [Background] Luckhaupt SE, Dahlhamer JM, Ward BW, Sweeney MH, Sestito JP, Calvert GM. Prevalence and work-relatedness of carpal tunnel syndrome in the working population, United States, 2010 National Health Interview Survey. Am J Ind Med. 2013 Jun;56(6):615-24. doi: 10.1002/ajim.22048. Epub 2012 Apr 11. PMID 22495886